CLINICAL TRIAL: NCT00522132
Title: Phase II Randomized, Double-Blind Study of the Efficacy, Safety, Tolerability, and Pharmacokinetics of Intravenous Artesunate in Children With Severe Malaria
Brief Title: Phase II Artesunate Study in Severe Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Severe Malaria in African Children Consortium (Other)
Responsible Party: Jörg J. Möhrle, Medicines for Malaria Venture
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDCTP/MMV07-01; EDCTP Grant #2004.01.M.d2
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Malaria
Keywords: intravenous artesunate; severe malaria; Plasmodium falciparum; Africa; Severe Plasmodium falciparum Malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artesunate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cohort 1 (Active Comparator): 2.4 mg/kg iv artesunate at 0, 12, 24, 48and 72 hours
  Interventions: Drug: Artesunate
- cohort 2 (Experimental): 4.0 mg/kg iv Artesunate at 0, 24 and 48 h
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — intravenous application

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of 2 intravenous artesunate dosing regimens (2.4 mg/kg initially and at 12, 24, 48, and 72 hours or 4.0 mg/kg initially and at 24 and 48 hours) in clearing P. falciparum parasites in children with severe malaria.

Secondary objectives include:

* To compare the tolerability and safety of the 2 intravenous artesunate dosing regimens.
* To evaluate differences in the pharmacokinetic profile of intravenous artesunate by patient age and clinical presentation.

DETAILED DESCRIPTION:
This is a Phase II, double-blind, multicenter, randomized, parallel-group study of the antimalarial activity and safety of 2 intravenous artesunate regimens in children with severe P. falciparum malaria (Appendix B). It will compare the efficacy, safety and tolerability of the SEAQUAMAT regimen, the recommended dosing regimen for adults,8 which requires twice daily artesunate dosing on the first day, to a simpler once daily regimen. The study will also evaluate the pharmacokinetic profile of artesunate in pediatric patients.

Prior to study initiation, the protocol will be approved by the Independent Ethics Committee/Institutional Review Board(s) (IEC/IRB) of each site and the national regulatory authority of each study site.

Approximately 200 patients will be randomized at 3 study sites in Africa, which are part of the Severe Malaria in African Children (SMAC) network. Patients will be randomized to 1 of 2 treatment cohorts:

* Cohort 1: artesunate 2.4 mg/kg initially, and at 12, 24, 48, and 72 hours (12 mg/kg total dose); or
* Cohort 2: artesunate 4 mg/kg initially, and at 24 and 48 hours (12 mg/kg total dose), normal saline will be administered as a placebo at 12 and 72 hours in order to maintain the study blind.

The study is divided into 3 main periods including the Pre-Treatment Period (Screening/Day 0), the Treatment Period (Days 0 through 3; Day 0 is the first day of study drug dosing), and the Post-Treatment Period (including evaluations on Days 7, 14, and 28). Children presenting to the study hospitals with signs/symptoms of severe malaria will be screened for study enrollment. Those with presumed severe malaria will be identified and informed consent for participation from parents/guardians will be obtained while confirmation of malaria is determined by microscopic analysis of a Giemsa-stained thick smear. Patients who meet study inclusion criteria and none of the exclusion criteria will be randomized and promptly treated with 1 of the artesunate regimens, while hospitalized for at least 4 days (Days 0, 1, 2, and 3). Adjunctive therapy, including fluids, glucose, and blood, will follow SMAC standards, based on WHO guidelines for the treatment of severe malaria (Appendix C). As soon as the patient is able to receive oral medication and no signs and symptoms of severe malaria are present, but not before the last pharmacokinetic sample is taken (approximately 50 hours after the start of therapy), a single dose of sulfadoxine/pyrimethamine will be administered to ensure parasitological cure. Patients who received sulfadoxine/pyrimethamine within 14 days prior Study Day 0 will receive mefloquine instead of SP,, to ensure effective parasitological cure.

If the parasitemia is controlled and the safety laboratory tests from Day 3 indicate no clinical concern warranting prolonged hospitalization, the patient may be discharged at the discretion of the investigator. If a patient is discharged from the hospital on Day 3, he/she will return to the study site on Day 7 for evaluation. If the patient is unable to tolerate oral liquids or food within 6-24 hours after the last dose of artesunate, the patient will continue to be hospitalized and treated with parenteral antimalarial therapy until he/she is able to resume oral intake or a total of 7 days of therapy have been completed. All patients will return to the study site for evaluation on Days 14 and 28 to assess resolution of clinical complications and monitor for safety of therapy.

Efficacy will be assessed by various parasite clearance parameters. Safety evaluations including physical examinations, vital signs, hematology and chemistry laboratory parameters and monitoring of adverse events will be performed throughout the study. Pharmacokinetic assessments will be performed at 3 different timepoints during the study.

If adverse events reported during the study are unresolved by Day 28, patients will be followed for an additional 30 days or until resolution of the event or determination that no further medical management is deemed necessary. Similarly, the investigator will instruct the parents/guardians to return the patient to the study site if any untoward event occurs within 30 days of completing study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children aged 6 months and ≥ 5kg to 10 years, inclusive.
* Clinical diagnosis of severe P. falciparum malaria (see Appendix B) requiring hospitalization.
* Parasitemia (more than 5,000 parasites/microL on initial blood smear).
* Availability of child's parent/guardian and their willingness to provide written informed consent in accordance to local practice.
* Willingness and ability to comply with the study protocol for the duration of the study.
* Willingness to remain in the hospital for 4 days

Exclusion Criteria:

* Known serious adverse reaction or hypersensitivity to artemisinins, including artesunate, artemether, dihydroartemisinins or Co-Artem (artemether/lumefantrine).
* Any underlying disease that may compromise the diagnosis and the evaluation of the response to the study medication (including concomitant infection, concomitant neurological disease and malnutrition)
* Participation in any investigational drug study during the 30 days prior to Screening.
* Adequate anti-malarial treatment within 24 hours prior to admission.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with parasite clearance (more than 99% reduction from the baseline asexual parasite count) at 24 hours after initiation of study drug. | 24 hours after initiation of study

SECONDARY OUTCOMES:
Time to total clearance of asexual parasites (PC100) | after study drug administration
Time to 99% reduction of asexual parasites (PC99) | after study drug administration
Time to 90% reduction of asexual parasites (PC90) | after study drug administration
PCR corrected Adequate Clinical and Parasitological Response on day 28 | on day 28
plasma concentrations of artesunate following intravenous administration | after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kremsner, MD, Principal Investigator — Universität Tübingen
Locations (3):
- Gabon (2):
  - Albert Schweitzer Hospital, Lambaréné
  - Universite de Medecine et Science de la Sante, Libreville
- Queen Elizabeth Central Hospital, Blantyre, Malawi

REFERENCES:
- [Derived] Kremsner PG, Taylor T, Issifou S, Kombila M, Chimalizeni Y, Kawaza K, Bouyou Akotet MK, Duscha M, Mordmuller B, Kosters K, Humberg A, Miller RS, Weina P, Duparc S, Mohrle J, Kun JF, Planche T, Teja-Isavadharm P, Simpson JA, Kohler C, Krishna S. A simplified intravenous artesunate regimen for severe malaria. J Infect Dis. 2012 Jan 15;205(2):312-9. doi: 10.1093/infdis/jir724. Epub 2011 Dec 15. PMID 22180622